CLINICAL TRIAL: NCT00886015
Title: Partnership for the Rapid Elimination of Trachoma (PRET) Clinical Trial of Evaluation of Modified Instrumentation for Surgery to Correct Trichiasis
Brief Title: Modified Instrumentation for Surgery to Correct Trichiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Emily Gower, Associate Professor of Ophthalmology, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00019216
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Trachoma
Keywords: Trachoma; trichiasis; bilamellar tarsal rotation procedure
MeSH Terms: conditions — Trachoma; Trichiasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TT Clamp (Experimental): The TT clamp will be used in trichiasis surgery.
  Interventions: Device: TT Clamp
- Standard BLTR Technique (Active Comparator): Standard BLTR technique will be used in trichiasis surgery.
  Interventions: Procedure: Standard BLTR Technique

INTERVENTIONS:
Device: TT Clamp — trichiasis surgery performed with TT clamp
  Arms: TT Clamp
Procedure: Standard BLTR Technique — bilamellar tarsal rotation procedure in trichiasis surgery
  Arms: Standard BLTR Technique

SUMMARY:
Trachoma, an ocular infection caused by C. trachomatis, is the second leading infectious cause of blindness worldwide. Years of repeated infection with C. trachomatis cause the eyelid to scar and contract and ultimately to rotate inward such that the eyelashes rub against the eyeball and abrade the cornea (trichiasis). The World Health Organization (WHO) has endorsed a multi-faceted strategy to combat trachoma which includes surgery to repair lids distorted by trachoma (trichiasis) in imminent danger of vision loss. Current evidence suggests that long-term success rates of trichiasis surgery are less than optimal due to variation in surgical technique. Previous research by this study team has demonstrated that shorter incisions have a higher rate of trichiasis recurrence. In addition, observations by this team's oculoplastic surgeon have led to the hypothesis that granuloma formation and lid contour abnormalities may result from current surgical practices. The objective of this study is to compare outcomes of trichiasis surgeries performed with the newly developed trachomatous trichiasis (TT) clamp versus surgeries following standard technique (bilamellar tarsal rotation procedure or BLTR).

DETAILED DESCRIPTION:
Field observations in 2005 by this study's PI and oculoplastic surgeon revealed some significant departures from current trichiasis surgery procedure (bilamellar tarsal rotation procedure or BTRP), as described in the WHO manual, "Trichiasis Surgery for Trachoma-the Bilamellar Tarsal Rotation Procedure". These procedural departures were felt to contribute to adverse outcomes, including trichiasis recurrence, granuloma formation and lid contour abnormalities. This study team developed a new surgical tool, the TT clamp, to help improve surgical outcomes following BLTR.

A randomized, single-masked clinical trial will be implemented in the Mtwara region in Tanzania. Study participants will be randomized on a 1:1 basis to surgery with the TT clamp or to surgery with standard BLTR equipment. All surgeries will take place at surgical centers in Mtwara and Lindi over an 8-month period.

Baseline assessment for severity of trichiasis and other predictors of surgical failure will be carried out prior to surgery. Follow-up is planned at 2 weeks (for suture removal), 6 weeks, 12 months, and 24 months post-surgery. At each follow-up visit participants will be assessed for evidence of unfavorable outcomes, including trichiasis recurrence, granuloma formation, and lid contour abnormalities. All outcomes will be assessed clinically by a trained observer who is masked to intervention status.

ELIGIBILITY:
Inclusion Criteria:

* Presence of upper lid trichiasis: defined by at least one eyelash touching the globe of the eye or evidence of epilation
* No previous report of trichiasis surgery in at least one eye with trichiasis:

  * eyes with prior surgery are already at high risk due to the prior surgery, and their inclusion may decrease our ability to clearly evaluate our primary outcome
  * if unilateral surgery has been performed previously, only the eye without prior history of surgery will be in the study, even if both eyes require surgery
* Age 18 or older (in order to provide consent as an adult): the vast majority of trichiasis patients are aged 18 or older
* At time of enrollment, subjects must state their intention to remain in the area for two years to facilitate study follow-up

Exclusion Criteria:

* Absence of upper lid trichiasis
* Prior trichiasis surgery on both eyes
* Age 18 or younger
* Subjects who are transiently in the area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1927 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Gower, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be provided to investigators through application to the data committee at Johns Hopkins University.

REFERENCES:
- [Derived] Gower EW, Munoz B, Rajak S, Habtamu E, West SK, Merbs SL, Harding JC, Alemayehu W, Callahan EK, Emerson PM, Gebre T, Burton MJ. Pre-operative trichiatic eyelash pattern predicts post-operative trachomatous trichiasis. PLoS Negl Trop Dis. 2019 Oct 7;13(10):e0007637. doi: 10.1371/journal.pntd.0007637. eCollection 2019 Oct. PMID 31589610
- [Derived] Gower EW, West SK, Harding JC, Cassard SD, Munoz BE, Othman MS, Kello AB, Merbs SL. Trachomatous trichiasis clamp vs standard bilamellar tarsal rotation instrumentation for trichiasis surgery: results of a randomized clinical trial. JAMA Ophthalmol. 2013 Mar;131(3):294-301. doi: 10.1001/jamaophthalmol.2013.910. PMID 23494035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-level eye screenings were conducted to identify all trichiasis cases in the community. Patients were scheduled for surgery. On the day of surgery they were invited to join the study if they were eligible.
Pre-assignment Details: 963 individuals assigned to Trachomatous Trichiasis (TT) clamp, 6 did not participate. 3 refused surgery, 2 ineligible because of lower eyelid trichiasis only, 1 participant did not present for surgery.
  964 individuals assigned to Standard, 4 did not participate. 2 refused surgery, 2 ineligible because of lower eyelid trichiasis only.
Groups:
- Standard Instrumentation: Eyelids operated with standard BLTR instrumentation
- TT Clamp: Eyelids operated with the TT clamp instead of standard BLTR instrumentation. The TT clamp replaces the 2 hemostats and lid plate
Period: Overall Study
Arm/Group | Standard Instrumentation | TT Clamp
Started | 1674 (1674 eyes; 960 participants) | 1671 (1671 eyes; 957 participants)
Completed | 1674 (1674 eyes; 960 participants) | 1669 (1669 eyes; 956 participants)
Not Completed | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: 1927 participants were originally enrolled. 10 participants did not undergo surgery for the following reasons: refused surgery (5), ineligible because of lower eyelid trichiasis only (4), or surgery was delayed and patient did not attend (1). The final total number of participants was 1917.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Instrumentation | TT Clamp | Total
Number analyzed (Participants) | 960 | 957 | 1917
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (13.1) | 54.9 (13.5) | 55.2 (13.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 722 | 705 | 1427
  Male | 238 | 252 | 490
Region of Enrollment [Number; unit: participants]
  Tanzania | 960 | 957 | 1917
Trichiasis [Number; unit: eyelids] — mild, moderate, severe
  eyelids
    mild | 347 | 303 | 650
    moderate | 453 | 423 | 876
    severe | 874 | 945 | 1819

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyelids With Presence of Recurrent Trichiasis
Description: Trichiasis: 1 or more eyelashes touching globe in primary position
Time Frame: 2 years
Population: Of the 1671 eyes initially assigned to TT Clamp, 1 participant (2 eyelids) was excluded from TT Clamp analysis because participant died before follow-up.
Measure: Number; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | TT Clamp | Standard BLTR Technique
Number analyzed (Participants) | 956 | 960
Number analyzed (eyelids) | 1669 | 1674
eyelids
  Normal | 948 | 1062
  TT Recurrence | 721 | 612
Statistical Analysis 1: Comparison: TT Clamp vs Standard BLTR Technique; Test type: Superiority or Other; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.96 to 1.93]

2. Primary Outcome: Number of Eyelids With Pyogenic Granuloma
Description: A pyogenic granuloma was defined as a sessile growth of 2 mm or more in diameter on the tarsal conjunctiva.
Time Frame: 2 years
Population: Of the original 1771 eyelids assigned to TT clamp, 1 participant (2 eyelids) was excluded from TT Clamp analysis because participant died before follow-up
Measure: Number; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | TT Clamp | Standard BLTR Technique
Number analyzed (Participants) | 956 | 960
Number analyzed (eyelids) | 1669 | 1674
eyelids
  Granuloma | 281 | 375
  Normal | 1388 | 1299
Statistical Analysis 1: Comparison: TT Clamp vs Standard BLTR Technique; Test type: Superiority or Other; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.46 to 0.98]

3. Primary Outcome: Number of Eyelids Experiencing an Unfavorable Outcome
Description: At least 1 unfavorable outcome, including mild, moderate, or severe trichiasis; granuloma; or mild, moderate, or severe eyelid contour abnormality
Time Frame: 2 years
Population: as for outcome 2
Measure: Number; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | TT Clamp | Standard BLTR Technique
Number analyzed (Participants) | 956 | 960
Number analyzed (eyelids) | 1669 | 1674
eyelids
  Any unfavorable outcome | 1017 | 1055
  Normal | 652 | 619
Statistical Analysis 1: Comparison: TT Clamp vs Standard BLTR Technique; Test type: Superiority or Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.66 to 1.18]

4. Primary Outcome: Number of Eyelids With Normal or Mild Eyelid Contour Abnormalities vs Moderate or Severe Eyelid Contour Abnormalities
Description: Eyelid contour abnormalities (ECA) were graded by photographs of the eyes. In the primary outcome measure, normal eyes and mild eyelid contour abnormalities are considered together, and moderate or severe eyelid contour abnormalities are considered together. ECA severity is defined as follows:
  Mild: Vertical deviation from the natural contour < 1 mm in height (less than half the pupil height in daylight) and affecting < 1/3 of horizontal eyelid length; Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length; Severe: Vertical deviation from the natural contour > 2 mm in height (more than the pupil height in daylight) or a defect > 2/3 of the horizontal eyelid length
Time Frame: 2 years
Population: as for outcome 2
Measure: Number; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | TT Clamp | Standard BLTR Technique
Number analyzed (Participants) | 956 | 960
Number analyzed (eyelids) | 1669 | 1674
eyelids
  No/Mild ECA | 1549 | 1500
  Moderate/Severe ECA | 120 | 174
Statistical Analysis 1: Comparison: TT Clamp vs Standard BLTR Technique; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.44 to 0.98]

5. Secondary Outcome: Number of Eyelids With Mild, Moderate, Severe, or no Eyelid Contour Abnormality
Description: Eyelid contour abnormalities (ECA) were graded by photographs of the eyes. ECA severity is defined as follows:
  Mild: Vertical deviation from the natural contour < 1 mm in height (less than half the pupil height in daylight) and affecting < 1/3 of horizontal eyelid length; Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length; Severe: Vertical deviation from the natural contour > 2 mm in height (more than the pupil height in daylight) or a defect > 2/3 of the horizontal eyelid length
Time Frame: 2 years
Population: Of the 1771 participants originally assigned to TT Clamp, 1 participant (2 eyelids) was excluded from TT Clamp analysis because participant died before follow-up
Measure: Number; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | TT Clamp | Standard BLTR Technique
Number analyzed (Participants) | 956 | 960
Number analyzed (eyelids) | 1669 | 1674
eyelids
  Normal | 1397 | 1278
  Mild ECA | 152 | 222
  Moderate ECA | 89 | 131
  Severe ECA | 31 | 43
Statistical Analysis 1: Comparison: TT Clamp vs Standard BLTR Technique; Mild ECA compared with Normal; Test type: Superiority or Other; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.42 to 0.97]
Statistical Analysis 2: Comparison: TT Clamp vs Standard BLTR Technique; Moderate ECA compared with Normal; Test type: Superiority or Other; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.39 to 1.01]
Statistical Analysis 3: Comparison: TT Clamp vs Standard BLTR Technique; Severe ECA compared with Normal; Test type: Superiority or Other; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.35 to 1.10]

6. Secondary Outcome: Number of Eyelids With Normal, Mild, Moderate, or Severe Trachomatous Trichiasis
Description: Trichiasis is generally defined as 1 or more eyelashes touching globe in primary position. Classifications of trichiasis severity are as follows:
  Mild: 1-4 Eyelashes touching globe, no epilation OR 1-10 Eyelashes epilated, no eyelashes touching globe; Moderate: 5-9 Eyelashes touching globe, no epilation OR 1-4 Eyelashes touching globe and 1-10 eyelashes epilated; Severe: 5-9 Eyelashes touching globe and 1-10 eyelashes epilated OR 10 Eyelashes touching globe, regardless of epilation status OR 11-20 Eyelashes epilated, regardless of eyelashes touching globe OR Entire eyelid epilated, regardless of eyelashes touching globe
Time Frame: 2 Years
Population: Of the 1669 TT eyelids and 1674 BLTR eyelids included in the initial analysis, 13 eyes (4 in the TT clamp group, 9 in the BLTR group) without TT at 1 year underwent operation between years 1 and 2. They are not included in the data for severity of recurrence because we do not know the TT severity.
Measure: Number; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | TT Clamp | Standard BLTR Technique
Number analyzed (Participants) | 954 | 956
Number analyzed (eyelids) | 1665 | 1665
eyelids
  Normal | 948 | 1062
  Mild TT Recurrence | 476 | 417
  Moderate TT Recurrence | 121 | 86
  Severe TT Recurrence | 120 | 100
Statistical Analysis 1: Comparison: TT Clamp vs Standard BLTR Technique; Test type: Superiority or Other; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.97 to 1.53]

ADVERSE EVENTS:
Time Frame: through 2 years
Arm/Group | Standard Instrumentation | TT Clamp
Serious Adverse Events (participants affected / at risk) | 0/960 | 0/957
Other Adverse Events (participants affected / at risk) | 15/960 | 12/957
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Instrumentation (N=960) | TT Clamp (N=957)
Excess intraoperative bleeding (Eye disorders) | 4 (4) | 0 (0)
Division of Eyelid Margin (Eye disorders) | 2 (2) | 0 (0)
postoperative bleeding (Eye disorders) | 5 (5) | 4 (4)
necrosis (Eye disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No